CLINICAL TRIAL: NCT03166878
Title: Phase I/II Study to Determine the Safety, Tolerability, Biological Activity and Efficacy of Universal CRISPR-Cas9 Gene-Editing CAR-T Cells Targeting CD19(UCART019) in Patients With Relapsed or Refractory CD19+ Leukemia and Lymphoma
Brief Title: A Study Evaluating UCART019 in Patients With Relapsed or Refractory CD19+ Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Molecular & Immunological Department, Bio-therapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-021
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: B Cell Leukemia; B Cell Lymphoma
Keywords: CAR-T; Cancer treatment; Immunotherapy; Adoptive cell therapy; Chimeric antigen receptor; Universal CAR-T
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (UCART019) (Experimental): The UCART019 will be administered by i.v. injection over 20-30 minutes as a using a "split dose" approach to dosing: Day 0: 10% of total dose. Day 1: 30% of total dose if patient is stable (no significant toxicity) from prior dose. D2: 60% of total dose if patient is stable (no significant toxicity) from prior dose
  Interventions: Biological: UCART019

INTERVENTIONS:
Biological: UCART019 — Day 0: 10% of total dose Day 1: 30% of total dose if patient is stable (no significant toxicity) from prior dose. D2: 60% of total dose if patient is stable (no significant toxicity) from prior dose

SUMMARY:
Autologous T cells engineered to express chimeric antigen receptors (CARs) against leukemia antigens such as CD19 on B cells have shown promising results for the treatment of relapsed or refractory B-cell malignancies. However, a subset of cancer patients especially heavily pretreated cancer patients could be unable to receive this highly active therapy because of failed expansion. Moreover, it is still a challenge to manufacture an effective therapeutic product for infant cancer patients due to their small blood volume. On the other hand, the inherent characters of autologous CAR-T cell therapy including personalized autologous T cell manufacturing and widely "distributed" approach result in the difficulty of industrialization of autologous CAR-T cell therapy. Universal CD19-specific CAR-T cell(UCART019),derived from one or more healthy unrelated donors but could avoid graft-versus-host-disease (GVHD) and minimize their immunogenicity, is undoubtedly an alternative option to address above-mentioned issues. We have generated gene-disrupted allogeneic CD19-directed BBζ CAR-T cells (termed UCART019) by combining the lentiviral delivery of CAR and CRISPR RNA electroporation to disrupt endogenous TCR and B2M genes simultaneously and will test whether it can evade host-mediated immunity and deliver antileukemic effects without GVHD.

The main goal of the phase 1 portion of this phase 1/2 trial is to evaluate the safety and tolerability of several doses of UCART019 in patients with relapsed or refractory CD19+ leukemia and lymphoma, so as to establish the recommended dose and/or schedule of UCART019 for phase 2 portion. The recommended Phase 2 dose will be defined as the highest dose level of UCART019 that induced DLT in fewer than 33% of patients (i.e., one dose level below that which induced DLT in at least two of six patients). Phase 2 portion of the trial will not be initiated until the recommended Phase 2 dose is determined. In the phase 2 portion of this trial, we will mainly determine if UCART019 help the body's immune system eliminate malignant B-cells. Safety of UCART019 and impact of this treatment on survival will also be observed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To evaluate the feasibility and safety of UCART019 in patients with relapsed or refractory CD19+ leukemia and lymphoma.
2. To evaluate the duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells. Real Time polymerase chain receptor (RT-PCR) analysis of peripheral blood(PB), bone marrow(BM) and lymph node will be used to detect and quantify survival of UCART019 over time.

SECONDARY OBJECTIVES:

1. For patients with detectable disease, measure anti-tumor response due to UCART019 cell infusions.
2. Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable UCART019 (loss of engraftment).

OUTLINE: This is a phase I, dose-escalation study of allogeneic CD19 CAR-T-cells followed by a phase II study.

The UCART019 will be administered by i.v. injection over 20-30 minutes as a using a "split dose" approach to dosing: 10% on day 0, 30% on day 1 and 60% on day 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant
2. 12 Years to 75 Years (Infant, Child, Adult, Senior)
3. Patient with relapsed or refractory CD19 positive B-cell leukemia or lymphoma
4. Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Adequate organ function

Exclusion Criteria:

1. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
2. Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis
3. Richter's syndrome
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
5. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
6. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
7. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
8. Patient has an investigational medicinal product within the last 30 days prior to screening
9. Previous treatment with investigational gene or cell therapy medicine products
10. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
11. Pregnant or nursing women

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety and Tolerability | 24 weeks
Highest dose of UCART019 that is estimated to result in defined DLT with the exception of allowable UCART019 infusion related 'expected' AEs, using CTCAE 4.0, in less than 1/3 patients | 8 weeks
Copy numbers of UCAR019 in PB, BM and lymph nodes | 24 weeks

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission.Descriptive statistics will be used | 24 weeks
Overall survival.Descriptive statistics will be used | 24 weeks
Progression free survival.Descriptive statistics will be used | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China